CLINICAL TRIAL: NCT02562430
Title: Neurobiological Underpinnings of Placebo Response in Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Cristina Cusin, MD, Staff Psychiatrist, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2014P000889
Record Dates: First submitted 2015-09-25; First posted 2015-09-29 (Estimated); Last update posted 2022-09-08 (Actual); Status verified 2022-09

CONDITIONS: Depression
Keywords: Placebo response
MeSH Terms: conditions — Depression | interventions — Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active Treatment (Experimental): 12.5 % will be randomized to Welbutrin XL in phase 1 of the study.
  Interventions: Drug: Welbutrin XL
- Placebo Group (Active Comparator): 87.5% will be randomized to receive placebo in phase 1 of the study.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Welbutrin XL — 12.5% of participants will receive Welbutrin XL in phase 1 of the study.
  Other Names: Buproprion XL
  Arms: Active Treatment
Drug: Placebo — 87.5% of subjects will be randomized to placebo in phase 1 of the study.
  Other Names: Sugar pill
  Arms: Placebo Group

SUMMARY:
In summary, the proposed research is novel with respect to design, technology, and its multi-level integration probing psychological and neurobiological constructs assumed to be crucially implicated in placebo response and has significant clinical and research implications for the future. Specifically, the future implications include: 1) identification of biomarkers and biosignatures of placebo responders, 2) new possibilities to understanding and manipulating the system, 3) possibly decreasing or eliminating a major confounder in clinical trials and drug development, and 4) refining treatments with novel drugs that decrease (in clinical trial) or increase (in clinical practice) the placebo response.

DETAILED DESCRIPTION:
The objective of this pilot study is to investigate possible dopaminergic mechanisms underlying the placebo response in MDD.

We expect that mesolimbic DA mechanisms implicated in reward anticipation, reinforcement learning, and expectation play a critical role in mediating placebo responses in MDD. A better understanding of the neurobiological basis of placebo has enormous potential on different levels. On a clinical level, the understanding of placebo mechanisms could lead to a number of applications for therapeutic purposes, such as developing drugs that could enhance the effects of a therapeutic relationship or accelerate the onset of action of an antidepressant by manipulating the placebo-related mechanisms, even if the patient is hopeless or severely anhedonic. On a level of clinical trial innovation, if we confirm the role of dopamine in placebo response and we comprehend how the placebo response mechanistically takes place, this could lead to developing new drugs that could block the placebo effects in clinical trial participants and greatly decrease if not eliminate the placebo effect nested even in those subject who are drug responders, therefore increasing the effect size and decreasing the sample size of studies. Moreover if we can identify biosignatures of placebo effect and use them to predict response, we could potentially enrich samples with subjects who are less likely to be placebo responders and again this would result in increased signal detection in a clinical trial. Finally, with this initial study we plan to lay the foundation for other studies to investigate how this dopaminergic circuitry is affected by other treatments, such as psychotherapy, and what are the changes that are similar or different between antidepressants, placebo and specific forms of psychotherapy, transcranial magnetic stimulation, electroconvulsive therapy or deep brain stimulation.

ELIGIBILITY:
Inclusion Criteria

In addition to fulfilling the diagnostic criteria for MDD, the following conditions must be met for patient eligibility:

1. Written informed consent
2. Men or women aged 18 to 60 years old
3. A score of 16 or greater on the Hamilton Depression Rating Scale -32 items (HAM-D- 32)
4. Continuing to meet criteria for current MDD at baseline and Clinical Global Impression Improvement (CGI) scores ≤ 3 (i.e. minimally improved or less) from the screen to the baseline visit
5. Only one failed one prior antidepressant in the current episode or are currently taking an antidepressant as defined by the MGH-ATRQ, in the current episode and are willing to take bupropion or placebo as augmentation, since we are using subjects as their own controls and we are comparing changes within subjects. Subjects with secondary anxiety disorders, like panic, GAD or simple phobia will be allowed, in order to make the population studied more representative of the general population of MDD.

Exclusion Criteria

1. Pregnant women or women of child bearing potential not using a medically accepted means of contraception.
2. Serious suicide or homicide risk.
3. Unstable medical illnesses, any history of seizure disorder.
4. The following DSM-IV diagnoses: a) organic mental disorders; b) substance use disorders, including alcohol abuse, within the last year; c) psychotic disorders; d) bipolar disorder; e) acute bereavement; f) severe borderline or antisocial personality disorder; g) history of eating disorder unless if in remission for ≥5 years prior to screening and presenting no current electrolyte abnormalities; h) current primary diagnoses of panic disorder, social phobia, PTSD, GAD, or OCD; i) mood congruent or mood incongruent psychotic features.
5. History of hepatic impairment or congestive heart failure.
6. Any history of abuse of stimulants or opiates.
7. Currently taking any exclusionary medications (i.e., antipsychotics, anticonvulsants, stimulants, dopaminergic agents), potential augmenting agents (e.g., T3, SAMe, St. John's Wort, lithium,). Gabapentin and pregabalin are allowed. Patients must have either no antidepressant treatment or stable (for at least 4 weeks prior to screening). No dose changes are allowed during the study. Monoamine oxidase inhibitors are excluded. Concomitant use of trazodone (up to 200 mg daily) is allowed. In agreement with patient's treating provider and under clinical monitoring, exclusionary drugs can be tapered and washed out prior to baseline visit.
8. Any investigational psychotropic drug within the last year.
9. Subjects who have not responded to two or more antidepressant trials of adequate doses (e.g., fluoxetine 40 mg/day or higher) and duration (e.g., ≥6 weeks) over the past five years according to the ATRQ.
10. History of inadequate response/poor tolerability to bupropion.
11. Subjects with medical contraindications to bupropion (e.g., history of seizures, uncontrolled electrolyte imbalance due to eating disorders, etc.) unless stable for 8 weeks prior to screening and there will be no changes during participation in the study.
12. Any unstable concomitant form of psychotherapy (depression-focused). Concomitant psychotherapy would be allowed if the frequency and the modality have been stable for the 8 weeks prior to screening and there will be no changes during the participation to the study
13. Receiving or have received during the index episode VNS, ECT or rTMS.
14. Color-blindness for blue or green (see fMRI task).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 73 (Actual)
Dates: Start 2016-08; Primary Completion 2022-08 (Actual); Study Completion 2022-08 (Actual)

PRIMARY OUTCOMES:
HAM-D 32 | 8 weeks

SECONDARY OUTCOMES:
Clinical Global Impressions | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Cusin, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Depression Clinical and Research Program at Massachusetts General Hospital, Boston, Massachusetts, United States